CLINICAL TRIAL: NCT04315792
Title: A Double-blind, Oral, Multiple-dose, Parallel, Randomized Study to Evaluate Efficacy and Safety of Endoxifen in Bipolar I Disorder Patients
Brief Title: Evaluate Efficacy and Safety of Endoxifen in Bipolar I Disorder Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jina Pharmaceuticals Inc. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry); Lambda Therapeutic Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0791-17
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Bipolar I Disorder
Keywords: Endoxifen, Bipolar I Disorder
MeSH Terms: interventions — 4-hydroxy-N-desmethyltamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoxifen Arm (Experimental): Endoxifen enteric-coated tablet (8 mg). Patients will continue treatment with their initial randomized medication for 3 weeks
  Interventions: Drug: Endoxifen
- Placebo Arm (Placebo Comparator): Placebo tablets of endoxifen. Patients will continue administration with their initial randomized medication for 3 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Endoxifen — Administration of Endoxifen for 3 weeks
  Arms: Endoxifen Arm
Drug: Placebo oral tablet — Administration of Placebo for 3 weeks
  Arms: Placebo Arm

SUMMARY:
The present study aims to evaluate the efficacy and safety of 8 mg endoxifen in the study population. As endoxifen represents a totally new class of drugs in the treatment of the bipolar disorder, it is essential to compare the drug against placebo to rule out the psychological influence upon study results. More so given the risks to patients and their communities from a medication whose efficacy has not been thoroughly evaluated against a placebo control. Thus, Endoxifen will be compared to placebo to demonstrate that the test product is active and to establish that the study is sufficiently sensitive to detect differences between the investigational products.

DETAILED DESCRIPTION:
Protein Kinase C (PKC) plays a major role in the regulation of both pre and postsynaptic neurotransmission. Excessive activation of PKC results in symptoms related to bipolar disorder. PKC exists as a family of closely related subspecies, has a heterogeneous distribution in the brain (with particularly high levels in presynaptic nerve terminals), and plays a crucial role in the regulation of neuronal excitability, neurotransmitter release, regulation of synaptic plasticity and various forms of learning and memory. Research findings show that the PKC pathway can be used as a target for developing treatment strategies for bipolar disorder. Endoxifen exhibited activity in inhibiting the PKC activity.

In patients with acute bipolar mania, rapid reduction of symptoms is a key treatment goal; however, there is also a need for effective maintenance of effect treatment beyond the period of acute stabilization. The current study will evaluate the efficacy and safety of Endoxifen in Bipolar I Disorder patients against a control placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, 18 to 65 (both inclusive) years of age willing to give written informed consent along with at least one first degree relative (the legally acceptable representative [LAR]) to participate in the study before initiating any study related procedures.
2. Patients must have a diagnosis of bipolar I disorder and currently display an acute manic episodes with or without mixed features according to DSM-5 criteria as judged by the Investigator.
3. Young Mania Rating Scale (YMRS) total score of > 20 and ≥4 on two of four core items (irritability, speech, content, disruptive/aggressive behavior) at screening and at randomization (baseline).
4. Score of >4 in Severity of illness criteria of Clinical Global Impressions- bipolar disorder (CGI-BP) Scale for overall illness at screening and at randomization (baseline).
5. Ready for voluntary hospitalization (along with the accompanying LAR if required and as advised by the Investigator) for the current manic episode 2 days prior to randomization up to 21 days of in-patient treatment period.
6. Last intake of the medication(s) for BPD should be 2-7 days prior to randomization depending upon the individual drug's plasma half-life.
7. Patient and / or LAR understand and agree to comply with all the study requirements.
8. Male patients of child begetting potential must be practicing adequate contraception.
9. Females of reproductive potential (which include girls who have entered puberty and all women who have a uterus and ovaries and have not completed menopause), must use anacceptable and effective method of avoiding pregnancy, starting at least four weeks before the first dose of study drug and continuing until at least one month after the last dose of study drug.
10. Subjects judged clinically not to be at serious suicide risk.

Exclusion Criteria:

1. Newly diagnosed patients and not having any suitable treatment exposure in the past for their bipolar mood disorder.
2. > 20% improvement in YMRS total scores between screening and randomization visits.
3. Patients who meet DSM-5 criteria for any psychiatric disorder other than Bipolar I Disorder with Acute Mania Episode with or without mixed features.
4. Patients with seizure disorder.
5. Obsessive compulsive disorder or any other co-morbid Axis I anxiety disorder
6. Patients with borderline or anti-social personality disorder of sufficient current severity to interfere with conduct of the study
7. Patients with classical premenopausal symptoms found at risk of developing intolerable hot flushes, irregular vaginal bleeding.
8. Use of the following medications:

   * Antihypertensive agents if stable dose has not been administered for at least 1 month before randomization
   * Antidepressants in the week (or a period of 5 half-lives of the drug) prior to randomization
   * Continuous daily or standing orders use of benzodiazepines during the month preceding screening (approximately 5 weeks prior to screening)
   * Potent cytochrome P450 (CYP) inducers and CYP2D6/CYP3A4 inhibitors 14 days prior to randomization
   * Depot antipsychotic medications within 1 dosing interval prior to randomization
   * Use of systemic estrogens 6 weeks prior to randomization
   * Patients currently on carbapenem agents
9. Any of the following laboratory abnormalities

   * Serum bilirubin ≥ 1.5 times ULN
   * Serum AST/ALT ≥ 2.5 times ULN
   * Serum TSH >10% above the ULN, regardless of treatment for hypothyroidism or hyperthyroidism
   * Serum triglyceride level > 2.5 times ULN
10. Patients with the following cardiac conditions are excluded:

    * Recent myocardial infarction (<12 months)
    * QTc prolongation (screening electrocardiogram with QTc >450 msec for men, QTc> 470 msec for women)
    * History of QTc prolongation or using concomitant medications (as judged by the Investigator) which prolong QTc interval
    * Sustained cardiac arrhythmia or history of sustained cardiac arrhythmia
    * De compensatory congestive heart failure
    * Complete left bundle branch block
    * First-degree heart block with PR interval > 0.22 seconds
11. Presence of a coagulation disorder; active or past history of venous thromboembolism including deep venous thrombosis or pulmonary embolism.
12. Current prolonged immobilization.
13. History or current presence of retinal pathology including retinal vein thrombosis
14. Increased risk of stroke as per the Investigator's discretion.
15. History of hypersensitivity or intolerance to tamoxifen or any other ingredients of the preparation.
16. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease as per history and medical examination.
17. Drug screen positive for any drug of abuse at screening (with the exception of benzodiazepines used in therapeutic dose for management of acute mania), active substance abuse in the past 2 months or history of substance dependence (excluding nicotine and caffeine) within 3 months of screening.
18. History of breast or uterine cancer, or abnormal uterine bleeding.
19. Current leukopenia or thrombocytopenia as judged by the Investigator in the best health interest of the subject.
20. Clinically significant suicidal or homicidal ideation.
21. Participation in a clinical trial of another investigational drug within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy and establish superiority of endoxifen 8 mg against placebo in Bipolar I Disorder patients (Mean change in total YMRS score) | 3 weeks
  Mean change in total YMRS score at Day 21 against baseline (in-patient setup)

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of all the treatments among Bipolar I Disorder patients (treatment related adverse events) | 3 weeks
  All treatment related adverse events including abnormal laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Treese, MD, Principal Investigator — Innovative Clinical Research, Inc.
Locations (1):
- 16420 NW 59 Avenue, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No